CLINICAL TRIAL: NCT01421927
Title: Safety of a Maintenance Therapy With Lenalidomide After Reduced-intensity Allogeneic Stem Cell Transplantation for Chemosensitive Relapsed Multiple Myeloma
Brief Title: Lenalidomide After Reduced-intensity Allogeneic Stem Cell Transplantation for Relapsed Multiple Myeloma
Acronym: REVALLO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/01
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Myeloma
Keywords: lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Start between Day+100 and Day+120 post-transplant
  - Initial dose: 5 mg/day every day
  In the absence of thrombocytopenia < 75000/mm3 or neutropenia < 1000/mm3 (with or without G-CSF), increase to the upper level than the ongoing one every third month up to the maximal dose of 15 mg/day every day.
  - Duration
  * until persistent stringent complete response for 3 months
  * or progression defined by IMWG criteria12
  * or unacceptable toxicity
  * or one year after transplant

SUMMARY:
Allogeneic stem cell transplantation (Allo-SCT) in multiple myeloma (MM) remains a controversial topic because of a high risk of relapse and a significant transplant-related mortality (TRM). In an effort to reduce the TRM, most allogeneic transplants in MM are now performed after reduced-intensity conditioning regimens. In these conditions, TRM usually range from 10 to 20%. However, reducing the intensity of the conditioning invariably increases the incidence of relapse to 45 to 60%. As a consequence, post-transplant strategies to reduce the incidence of relapse after reduced-intensity Allo-SCT should be considered and evaluated.

DETAILED DESCRIPTION:
Lenalidomide has a significant clinical activity in patients with relapsed or refractory MM and in patients relapsing after Allo-SCT. The mechanisms of action involve immunomodulation, anti-angiogenesis activity, direct anti tumor activity and effects on microenvironment. So far, the experience with lenalidomide after Allo-SCT has been limited to patients with progressive disease. In such patients, some responses are observed but most of them are transient with median progression-free survivals of less than one year. Lenalidomide used as maintenance therapy in patients with persistent rather than progressive disease might be a better approach.

Lenalidomide is interesting in the Allo-SCT setting also because some recent studies focusing on its immunological properties have suggested that the molecule could stimulate the graft versus myeloma effect. First, it has been demonstrated in vitro that lenalidomide can inhibit the proliferation and the suppressor function of regulatory T cells. Secondly, a clinical study using lenalidomide as salvage therapy after Allo-SCT demonstrated an increase of activated T cells and NK cells. Finally, a case report described a patient's response to lenalidomide associated with the development of an acute graft versus host disease.

Taken together, these data suggest that patients with MM who have a persistent disease after a reduced-intensity Allo-SCT might benefit from a post-transplant maintenance strategy with lenalidomide by a direct anti-tumor effect and a stimulation of the graft versus myeloma effect. The primary objective of this study is to evaluate the safety of such a strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years
* Multiple Myeloma in 2nd or 3rd complete or partial response*
* Disease never refractory to lenalidomide
* Lenalidomide treatment ≤ 9 months
* HLA related or unrelated donor (matched 10/10 or mismatched 9/10 HLA-C high resolution level or HLA-DQ high or low resolution level)
* Insured under Social Security
* Information and consent signed

Exclusion Criteria:

* Stable or progressive disease
* Hypersensitivity to lenalidomide or excipients
* Lenalidomide treatment > 9 months
* Absence of efficient contraception in women or men
* Cardiac insufficiency (ejection fraction < 50% by echocardiography)
* Pulmonary disease characterized by DLCO < 60%
* Severe renal insufficiency (clearance of creatinin < 30 ml/min)
* Hepatic disease characterized by ASAT and/or ALAT and/or total bilirubin > 2 times the upper normal value except in case of Gilbert's disease
* Bacterial, Viral or Fungal uncontrolled infections
* No contraceptive method for Female subjects of childbearing potential
* No use of condoms for males subjects
* Pregnant or breast feeding woman
* History of previous cancer (other than myeloma) except if the patient is in complete remission for more than 5 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety of lenalidomide | 1 year
  The main judgement criteria will be the occurrence of adverse events (AE) requiring the definitive interruption of lenalidomide :
  * Grade 3 or 4 adverse event according to the Common Terminology Criteria for Adverse Events (CTCAE) v3.0 occurring at the lowest dose of lenalidomide or
  * Steroid-refractory acute (Seattle criteria) or chronic (National Institutes of Health (NIH) criteria) graft versus host disease or
  * Transplant-related death

SECONDARY OUTCOMES:
One-year Progression-Free Survival | one year
  Progression defined according to International Myeloma Working Group (IMWG) criteria
One-year Overall Survival | one year
  all-cause death
One-year Transplant Related Mortality | one year
One-year incidence of Relapse/Progression | one year
  Progression defined according to IMWG criteria
Incidences of acute and chronic Graft versus Host Disease | one year
  Acute graft versus host disease according to Seattle criteria. Chronic graft versus host disease according to NIH criteria.
Immunophenotypic analysis of blood B, T, NK and dendritic cells | one year
Chimerism analysis | one year
safety of lenalidomide | one year
  all adverse events, graded according to NCI-CTCAE v3

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Vigouroux, Dr, Principal Investigator — University Hospital, Bordeaux; Adélaïde DOUSSAU, Dr, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU Bordeaux - Hôpital Haut-Lévêque, Pessac, France